CLINICAL TRIAL: NCT05374954
Title: Safety and Immunogenicity Study on Omicron Inactivated COVID-19 Vaccine and Prototype Inactivated COVID-19 Vaccine in Population Aged 18 Years Old and Above Vaccinated the Prototype Inactivated COVID-19 Vaccine
Brief Title: Study on Sequential Immunization of Omicron Inactivated COVID-19 Vaccine and Prototype Inactivated COVID-19 Vaccine in Population Aged 18 Years Old and Above
Acronym: COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Hunan Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CNBG-BIBP-O-2022004
Record Dates: First submitted 2022-05-13; First posted 2022-05-16 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: COVID-19; vaccine; inactivated vaccine
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (28):
- A1：one dose, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive one dose from 3 months to 6 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- A2：one dose, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive one dose from 3 months to 6 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- A3：one dose, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive one dose from 6 months to 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- A4：one dose, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive one dose from 6 months to 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- B1：one dose, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive one dose from 3 months to 6 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- B2：one dose, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive one dose from 3 months to 6 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- B3：one dose, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive one dose from 6 months to 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- B4：one dose, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive one dose from 6 months to 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- C1：two doses, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- C2：two doses, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- C3：two doses, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- C4：two doses, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- C5：two doses, 18-59 years old, more than 12 months after 2 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart more than 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- C6：two doses, 18-59 years old, more than 12 months after 2 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart more than 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- D1：two doses, 60 years old and above, from 3 months to 6 months after 2 doses of vaccination (Experimental): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- D2：two doses, 60 years old and above, from 3 months to 6 months after 2 doses of vaccination (Active Comparator): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- D3：two doses, 60 years old and above, from 6 months to 12 months after 2 doses of vaccination (Experimental): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- D4：two doses, 60 years old and above, from 6 months to 12 months after 2 doses of vaccination (Active Comparator): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 2 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- E1：two doses, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- E2：two doses, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- E3：two doses, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- E4：two doses, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- E5：two doses, 18-59 years old, more than 12 months after 3 doses of vaccination (Experimental): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart more than 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- E6：two doses, 18-59 years old, more than 12 months after 3 doses of vaccination (Active Comparator): subjects aged 18-59 years old will be blinded and receive two doses of vaccine with 28 days apart more than 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- F1：two doses, 60 years old and above, from 3 months to 6 months after 3 doses of vaccination (Experimental): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- F2：two doses, 60 years old and above, from 3 months to 6 months after 3 doses of vaccination (Active Comparator): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 3 months to 6 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- F3：two doses, 60 years old and above, from 6 months to 12 months after 3 doses of vaccination (Experimental): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- F4：two doses, 60 years old and above, from 6 months to 12 months after 3 doses of vaccination (Active Comparator): subjects aged 60 years old and above will be blinded and receive two doses of vaccine with 28 days apart from 6 months to 12 months after 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated — intramuscular injection in the deltoid muscle
  Arms: A1：one dose, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination; A3：one dose, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination; B1：one dose, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination; B3：one dose, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination; C1：two doses, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination; C3：two doses, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination; C5：two doses, 18-59 years old, more than 12 months after 2 doses of vaccination; D1：two doses, 60 years old and above, from 3 months to 6 months after 2 doses of vaccination; D3：two doses, 60 years old and above, from 6 months to 12 months after 2 doses of vaccination; E1：two doses, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination; E3：two doses, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination; E5：two doses, 18-59 years old, more than 12 months after 3 doses of vaccination; F1：two doses, 60 years old and above, from 3 months to 6 months after 3 doses of vaccination; F3：two doses, 60 years old and above, from 6 months to 12 months after 3 doses of vaccination
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — intramuscular injection in the deltoid muscle
  Arms: A2：one dose, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination; A4：one dose, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination; B2：one dose, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination; B4：one dose, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination; C2：two doses, 18-59 years old, from 3 months to 6 months after 2 doses of vaccination; C4：two doses, 18-59 years old, from 6 months to 12 months after 2 doses of vaccination; C6：two doses, 18-59 years old, more than 12 months after 2 doses of vaccination; D2：two doses, 60 years old and above, from 3 months to 6 months after 2 doses of vaccination; D4：two doses, 60 years old and above, from 6 months to 12 months after 2 doses of vaccination; E2：two doses, 18-59 years old, from 3 months to 6 months after 3 doses of vaccination; E4：two doses, 18-59 years old, from 6 months to 12 months after 3 doses of vaccination; E6：two doses, 18-59 years old, more than 12 months after 3 doses of vaccination; F2：two doses, 60 years old and above, from 3 months to 6 months after 3 doses of vaccination; F4：two doses, 60 years old and above, from 6 months to 12 months after 3 doses of vaccination

SUMMARY:
This is a randomized, double blind, positive controlled study to evaluate the safety and immunogenicity of Omicron COVID-19 Vaccine (Vero Cell), Inactivated in population aged 18 years old and above who have been vaccinated with 2 or 3 doses of COVID-19 Vaccine (Vero Cell), Inactivated manufactured by Beijing Institute of Biological Products, Co., Ltd.

DETAILED DESCRIPTION:
This is a randomized, double blind, positive controlled study to evaluate the safety and immunogenicity of Omicron COVID-19 Vaccine (Vero Cell), Inactivated in population aged 18 years old and above who have been vaccinated with 2 or 3 doses of COVID-19 Vaccine (Vero Cell), Inactivated manufactured by Beijing Institute of Biological Products, Co., Ltd. According to subject's age (18-59 vs 60 and above), doses of vaccination history ( 2 doses vs 3 doses), and vaccination interval, the subjects will be stratified and assigned randomly to the study groups ( Omicron inactivated COVID-19 Vaccine) or the control groups ( Prototype inactivated COVID-19 Vaccine) in a 2:1 ratio. All subjects will receive single dose or two doses of vaccine with a interval of 28 days. The occurrence of adverse events within 28 days and serious adverse events within 12 months after vaccination will be observed. The serum antibody levels, cellular immune responses will be analyzed at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 years old and above.
* By asking for medical history and physical examination, the investigator judged that the health condition is well.
* Has been vaccinated 2 or 3 doses of inactivated COVID-19 vaccine manufactured by BIBP more than 3 months.
* Female subjects of childbearing age are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 12 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* During the whole follow-up period of the study, be able and willing to complete the whole prescribed study plan.
* With self-ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Confirmed or suspected cases of SARS-CoV-2 Infection.
* Has a history of SARS, MERS, SARS-CoV-2 infection (self-report, on-site inquiry).
* Received one dose or more than 3 doses of inactivated COVID-19 vaccine manufactured by BIBP
* Received COVID-19 vaccine manufactured bu other companies (include mRNA, recombinant protein vaccines, vector vaccines, inactivated vaccines, etc.)
* Axillary body temperature > 37.3 ℃ before vaccination
* Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of inactivated SARS-CoV-2 vaccine have occurred (self-report, on-site inquiry).
* History of hospital-diagnosed thrombocytopenia or other coagulation disorder
* Known immunological impairment or low level with hospital diagnosis
* History of uncontrolled epilepsy, other progressive neurological disorders, or Guillain-Barre syndrome (self-report, on-site inquiry).
* Known or suspected concomitant serious diseases include: respiratory disease, acute infection or active chronic disease, liver and kidney disease, severe diabetes, malignant tumor, infection or allergic skin disease, HIV infection.
* Severe cardiovascular disease (cardiopulmonary failure, uncontrolled hypertension, etc.) diagnosed by the hospital, active chronic respiratory disease
* Received live attenuated vaccine within 1 month before enrollment.
* Received other vaccines within 14 days before enrollment.
* Be participating in or plan to participate in other vaccine clinical trials during this study.
* Contraindications related to vaccination as considered by other investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4200 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
The Geometric Mean Titer (GMT) of neutralizing antibody against Omicron SARS-CoV-2 | On Day 28 after vaccination
The four-fold increase rate of neutralizing antibody against Omicron SARS-CoV-2 | On Day 28 after vaccination
Incidence of adverse reactions | within 28 days after vaccination

SECONDARY OUTCOMES:
The GMT of neutralizing antibody against Omicron SARS-CoV-2 | On Day 14 after vaccination
The four-fold increase rate of neutralizing antibody against Omicron SARS-CoV-2 | On Day 14 after vaccination
Specific cellular immune response | within 28 days after vaccination
The neutralizing antibody GMT | on 3rd month, 6th month, 9th month, and 12th month after vaccination
The proportion of subjects with neutralizing antibody GMT ≥1:16，≥1:32 and ≥1:64 | on 3rd month, 6th month, 9th month, and 12th month after vaccination
The incidence of any adverse reactions/events | 28 days after each immunization
The incidence of serious adverse events (SAE) and adverse events special interest (AESI) | From the beginning of the first dose to 12 months after vaccination

OTHER OUTCOMES:
The neutralizing antibody GMT to different variants of SARS-CoV-2 | On Day 28 after vaccination
The IgG antibody lever against Omicron SARS-CoV-2 | On Day 14 and Day 28 after vaccination
The incidence of COVID-19 cases , including severe cases and deaths accompanied by COVID-19 | From 14 day after vaccination

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Linli County Center for Disease Control and Prevention, Changde, Hunan
  - Changning Center for Disease Control and Prevention, Changning, Hunan
  - Ningxiang Center for Disease Control and Prevention, Changsha, Hunan
  - Outpatient Department of Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan
  - Loudi Public Health Hospital, Loudi, Hunan
  - Xiangtan Center for Disease Control and Prevention, Xiangtan, Hunan
  - Luxi County Center for Disease Control and Prevention, Xiangxi, Hunan
  - Xiangxiang Center for Disease Control and Prevention, Xiangxiang, Hunan
  - Huarong County Center for Disease Control and Prevention, Yueyang, Hunan
  - You County Center for Disease Control and Prevention, Zhuzhou, Hunan

IPD SHARING:
Plan to Share IPD: No